CLINICAL TRIAL: NCT04715971
Title: Urinary Retention on an Acute Geriatric Hospitalisation Unit: Prevalence, Risk Factors and the Role of Screening, an Observational Cohort Study
Brief Title: Urinary Retention on an Acute Geriatric Hospitalisation Unit.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Katleen Fagard, Head of Clinic, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: mp08305
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Urinary Retention; Aged
Keywords: urinary retention; post-void residual volume; bladder scan; prevalence; risk factors; elderly
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted ≤72 hours to an acute geriatric hospitalisation unit.: All patients aged ≥75 years, admitted to the acute geriatric hospitalisation units of the University Hospitals Leuven in Belgium, were consecutively screened for inclusion within 72 hours of admission in a 2 month period (between October 26 and December 18, 2015).
  Interventions: Diagnostic Test: portable ultrasound bladder scan

INTERVENTIONS:
Diagnostic Test: portable ultrasound bladder scan — A post-void residual volume was measured using a Verathon BladdersScan BVI 3000.

SUMMARY:
Aim: The aim of this observational cohort study was to measure the prevalence of UR in patients aged ≥75 years on admission to an acute geriatric hospitalisation unit and to determine which at risk group would benefit from screening.

Methods: Post-void residual volumes (PVR) were measured within 3 days of admission with an ultrasound bladder scan. Uni- and multivariable analysis were used to determine risk factors associated with PVR ≥150 and ≥300 millilitres.

DETAILED DESCRIPTION:
1. Sample and setting An observational cross-sectional cohort study was conducted on the acute geriatric hospitalisation units of the University Hospitals Leuven in Belgium which have a collective capacity of 80 beds. All patients aged 75 years or older admitted with or without an indwelling urinary catheter between October 26 and December 18, 2015 were consecutively screened for inclusion within 72 hours of admission. Patients with urinary catheters for any other reason than UR, patients with ascites, dialysis, uro- or nephrostomy, terminally ill patients, and postoperative patients were not eligible for inclusion. Patients who refused to participate, who were unable to understand and carry out the instructions for the PVR measurement, with a urinary catheter for chronic UR, who were discharged or died during the inclusion process were excluded. The study was approved by the Ethics Committee Research of the University Hospitals Leuven (mp08305). The study nurse (SV) obtained a written informed consent from all patients who agreed to participate in the study, or from a proxy when the patient was incapable to provide written informed consent.
2. Procedures Prior to the start of the study, information sessions were organised for the nurses from the acute geriatric hospitalisation units, in which the study nurse (SV) explained the aim of the study and the data collection procedure. In addition, information was given on the use of the portable ultrasound bladder scan and the execution of a bladder scan.

   The nurses were asked to perform 3 consecutive post-void bladder scans as soon as possible after admission and at the latest within 72 hours of admission as standard of care during the study period. The highest value of the 3 consecutive PVR measurements was recorded. The study nurse (SV) was present on Monday, Wednesday and Friday morning, performed informed consents and performed bladder scanning in patients where this had not yet been done. Before performing the bladder scan, the patients were asked to urinate. Whenever possible, patients had to walk to the toilet in the bathroom, with or without assistance, meanwhile their mobility was assessed.

   Consecutively, the study nurse performed a bedside assessment. A mini-cog examination was performed and urinary symptoms, defaecation habits, and fall history were assessed by patient or caregiver interview using a structured questionnaire (SV). The demographic and remaining clinical data were collected from the patient's electronic medical records (SV, KH, KF).
3. Variables Outcome variables The PVR was measured using a portable ultrasound bladder scan (Verathon BladdersScan BVI 3000). Jalbani et al. found a high correlation (r²=0.97) between urinary catheterisation (gold standard) and bladder scanning and concluded that the use of the Verathon BladderScan BVI 3000 is as accurate as urinary catheterisations for measuring the PVR. As there are no official definitions or guidelines on what is considered a relevant PVR for UR, in this study we defined UR as a PVR of ≥150 millilitres. In addition, we also included a PVR ≥300 ml as secondary outcome. The cut-offs were chosen for the following reasons: the first bladder-filling sensation is felt at a volume of 150 ml. At a volume of 300 ml, the pressure receptors in the bladder wall will be activated, which creates a sense of fullness of the bladder and a need to urinate. Moreover, in clinical practice a PVR ≥300ml is often considered as threshold for insertion of a urinary catheter.

   Demographics The following patient characteristics were recorded: age, gender and living situation. Patients living alone at home and together at home were considered as living at home and patients living in an assisted living facility or nursing home were considered as not living at home. Patients living in a convent were considered as not living at home when they were functionally or cognitively impaired.

   Comorbidities Various comorbidities were retrospectively retrieved from the patient's electronic medical records: neurological, gynaecological and urological history, a history of diabetes type 1 or 2, recurrent falls (more than 1 fall episode in the last 6 months), and chronic kidney disease (CKD). CKD was defined as a glomerular filtration rate (eGFR, calculated using the CKD-EPI formula) of <60 ml/min/1.73 m². An age adjusted definition (<45 ml/min/1.73 m²) was also considered.

   Clinical evaluation Urinary incontinence was assessed by means of 3 questions: Do you have/does the patient have (1) an urge to urinate and involuntary loss of urine before reaching the toilet? (2) involuntary loss of urine when sneezing, coughing, lifting or moving something? (3) loss of small amounts or drops of urine without urge to urinate or loss of small drops of urine when changing position. Answering positive on these questions was classified as urge, stress or overflow incontinence, respectively. Dysuria was questioned as having a burning sensation or pain when urinating. Urinary frequency was questioned as urinating more often than usual. Voiding difficulty was questioned as straining to void. Subtotal voiding was questioned as the feeling of incomplete bladder emptying. Hypogastric pain was questioned as pain in the lower abdomen.

   Constipation was defined as the absence of stools for 3 or more days before the PVR measurement, or if patients reported having had less than 3 stools in the last week with a need to strain and mostly hard or lumpy stools, or if the patient had faecal impaction. Faecal impaction was defined as a large mass of compacted faeces in the rectum or colon on clinical or radiographical examination, that could not be spontaneously evacuated.

   The cognitive status of the patients was evaluated using the Mini-Cog. The Mini-Cog is a brief cognitive test that involves an assessment of an older person's ability to memorise three words, to draw a clock, and to recall the three words. Repeating only 1 or 2 of the 3 words and being unable to draw a clock correctly or not being able to repeat any of the words was considered as cognitive impairment.

   Mobility was assessed by walking to the bathroom and going to the toilet. All patients were asked to urinate on the toilet prior to the PVR measurements. Patients were considered mobile if they could walk back and forth to the toilet and if they were able to stand up from the toilet independently. The use of mechanical aids was permitted. Needing assistance from another person or not being able to walk was defined as impaired mobility.

   Laboratory evaluation and urinalysis The patient's renal function was evaluated by serum creatinine level and eGFR (calculated using the CKD-EPI formula).

   A urinary dipstick test was performed in all patients. In patients with positive leucocyte esterase or positive nitrites on the dipstick test, further urinalysis was performed. An automated leucocyte count of ≥10 leukocytes/mm³ and significant microscopic bacteriuria of >100.000 CFU/ml for which antibiotics were started by the treating physician was considered as UTI in this study. If the patient was taking antibiotics at the time of the urine sample and cultures remained negative, the presence of UTI was determined based on the leucocyte count.

   Medication For each patient the anticholinergic burden scale (ACB) score was calculated taking into account medication use in the last 24 hours before the PVR measurement. Individual drugs with high anticholinergic properties (ACB score ≥2), such as antipsychotics, antidepressants, as well as detrusor relaxants, were examined separately for their associations with UR. Antiepileptics, histamine H1 receptor antagonists, anti-diarrhoea medications, decongestive drugs, spasmolytics, muscle relaxants, and antiparkinsonian agents with ACB scores ≥2 were not considered individually. Low prevalence of these drugs prohibited statistical analysis.

   Reason for referral to the hospital The reasons for referral to the hospital were divided into the following categories: confusion, falls or immobility, urinary symptoms, cardiopulmonary symptoms, digestive symptoms, fever or non-specific symptoms with biochemical inflammation (elevated leucocytosis and elevated C-reactive protein) on admission, other. In patients with multiple reasons for admission, each reason was scored separately.
4. Statistical analysis Descriptive and comparative statistics were used. Normally distributed continuous variables were reported as means with standard deviations (SD). Not normally distributed continuous variables were reported as medians with interquartile ranges (IQR). Categorical variables were reported as numbers and percentages. Baseline characteristics and clinical variables of patients with a PVR of <150 ml versus ≥150 ml and a PVR of <300 ml versus ≥300 ml were compared using unpaired t-tests for normally distributed continuous variables. Pearson Chi-squared tests or Fisher's exact tests (if ≥1 cell had an expected count of less than 5) were used for dichotomous or nominal variables, and Mann-Whitney U tests for not normally distributed continuous variables or ordinal variables. All tests were 2-tailed, assuming a 5% significance level. Multivariable logistic regression models were used to determine independent predictors for a PVR ≥150 ml and a PVR ≥300 ml. Significant variables in the univariable analysis were considered in a forward stepwise logistic regression procedure. P-values (Likelihood ratios), odds ratios (OR), and 95% confidence intervals (CI) are reported. The software package used was SPSS version 20 (SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 75 years or older
* with or without a urinary catheter
* admitted no more than 72 hours to an acute geriatric hospitalisation unit of the Leuven University Hospitals

Exclusion Criteria:

* indwelling urinary catheter for another reason than acute urinary retention
* ascites
* dialysis
* uro- or nephrostomy
* terminally ill
* postoperative
* refusal to participate
* unable to understand and carry out the instructions for the post-void residual volume measurement

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 75 years or older on admission to an acute geriatric hospitalisation unit.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
post-void residual volume | measurement within 72 hours of admission to the acute geriatric hospitalisation unit
  residual volume after urinating measured with a portable ultrasound bladder scan (Verathon BladdersScan BVI 3000)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Flamaing, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Data are stored on a central secured server for data storage of the University Hospitals Leuven and are available upon contacting the corresponding author after publication, unless the journal asks for publication of the data on a datasharing site.